CLINICAL TRIAL: NCT01739374
Title: Phase 2-3 Study of Efficacy and Safety of Reduced Pelvic Floor Mesh Implants
Brief Title: Efficacy and Safety of Reduced Pelvic Floor Mesh Implants
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Principal Investigator, menahem neuman, Primary Investigator, Western Galilee Hospital-Nahariya
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HTA5969; 24411 (Other: Local IRB)
Record Dates: First submitted 2012-11-22; First posted 2012-12-03 (Estimated); Last update posted 2015-06-18 (Estimated); Status verified 2015-06

CONDITIONS: Post Operative Pain; Complication of Surgical Procedure
Keywords: pelvic floor reconstruction; mesh implants
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Device - Reduced mesh implants (Experimental): Patients treated with reduced mesh implants for POP reconstruction
  Interventions: Other: reduced mesh implants

INTERVENTIONS:
Other: reduced mesh implants — mesh for pelvic floor reinforcement

SUMMARY:
Pelvic organ prolapse is an herniation process, needing a mesh reconstruction for long lasting therapeutic effect. Yet, mesh implants were reported to be related to severe adverse effects. This study looks at the potential benefit of mesh size reduction regarding avoiding operative complications.

DETAILED DESCRIPTION:
Pelvic organ prolapse is a common disorder that results in significant patient morbidity. Approximately 1 in 9 women undergo surgery for the correction of pelvic organ prolapse (POP) and associated bladder and bowel dysfunction. Despite its common occurrence, the cause of POP remains largely unknown. Prolapse is thought to be caused by direct injury to the levator ani (LA) muscle, denervation of the pelvic floor musculature, or fascial damage incurred during childbirth trauma.

It is evident that pelvic organ prolapse (POP) occurs when the supporting pelvic floor becomes weakened or stretched, usually caused by childbirth, leading to descent of the pelvic organs to the vagina and beyond. This contributes to the impairment of pelvic organ function and a deterioration of patient quality of life. POP is estimated to severely affect approximately 11% of the female population.

Symptomatic POP patients might benefit from conservative management, such as the use of physiotherapy or vaginal pessaries. However, advanced POP necessitates surgical reconstruction. This might be achieved by the abdominal approach by an open operation or by laparoscopy, or by the vaginal approach. Synthetic permanent or absorbable meshes or biological grafts, or any synthesis of these might be used for reinforcement of the weakened pelvic floor structures that led to POP.

The need for reinforcement of the weakened fascia for achieving a long lasting cure of herniation processes is un-questionable. Given that the underlying pathology leading to POP is actually just a hernia of the pelvic floor, one must admit that the very same surgical principles used for any hernia repair are applicable for POP.

Most of the adverse effects are related to excessive implanted mesh mass. Thus, our goal with this study is to look at the issue of reducing the mesh size, surface area and the total mesh mass, assuming that the less quantity of left over implant the less mesh related complication will occur. The narrative for that is the notion that the natural pelvic floor connective tissue architecture is ligamentary and not "sheath like", while available pre-cut meshes are much too wide spread. This study concept is that reducing the mesh surface will lead to reduction with the mesh related complication. Given that the mesh implant size will be reduced, so will also be the wide of the extent of preliminary dissection, necessary for proper mesh placement. Thus, the dissection related adverse effects are expected to reduce as well.

ELIGIBILITY:
Inclusion Criteria:

-Patients with advanced pelvic organ prolapse

Exclusion Criteria:

- Patients with active infections or after pelvic irradiation

Ages: 35 Years to 95 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-05; Primary Completion 2014-05 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Intra-operative and post operative adverse effects | One year post operative
  Vaginal and pelvic pain upon VAS, vaginal mesh exposure, infections.

SECONDARY OUTCOMES:
Efficacy | One year
  Pelvic organ prolapse reconstruction upon the International Continence Society Pelvic Organ Prolapse Quantification System measurements

CONTACTS AND LOCATIONS:
Overall Officials: Menahem Neuman, Prof., Principal Investigator — Faculty of Medicine, Bar-Ilan Univ., Zafed
Locations (2):
- Israel (2):
  - Western Galilee MC, Nahariya
  - Ob-Gyn Dep., Western Galilee MC, Nahariya